CLINICAL TRIAL: NCT00630929
Title: A Study of the Efficacy and Tolerability of Once Daily Celebrex (Celecoxib) and Three Times Daily Ibuprofen vs. Placebo in the Treatment of Subjects With Osteoarthritis of the Knee
Brief Title: Efficacy and Safety of Celecoxib Versus Ibuprofen in the Treatment of Osteoarthritis of the Knee (Europe)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3191062
Record Dates: First submitted 2008-02-28; First posted 2008-03-07 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Ibuprofen; Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Active Comparator)
  Interventions: Drug: Ibuprofen
- C (Placebo Comparator)
  Interventions: Drug: Placebo
- B (Experimental)
  Interventions: Drug: Celecoxib

INTERVENTIONS:
Drug: Ibuprofen — 800 mg oral tablet 3 times daily with meals for 6 weeks
  Arms: A
Drug: Placebo — Matched placebo orally for 6 weeks
  Arms: C
Drug: Celecoxib — 200 mg oral capsule once daily with morning meal for 6 weeks
  Arms: B

SUMMARY:
To compare the efficacy and safety of celecoxib versus ibuprofen in subjects with osteoarthritis (OA) of the knee.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria:

* Aged >=40 years old
* Diagnosed with OA of the knee according to the American College of Rheumatology and OA in flare state at baseline visit
* Functional capacity class of I-III

Exclusion Criteria:

Exclusion criteria:

* Inflammatory arthritis or gout or pseudo-gout with acute flare within the past 2 years (subjects with fibrositis or fibromyalgia will not be excluded)
* Acute joint trauma at index joint within the past 3 months with active symptoms
* Score of >=20 on PHQ-9 or score of >=1 on PHQ-9 item i
* Use of mobility assisting device for <6 weeks or use of walker

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 388 (Actual)
Dates: Start 2003-01; Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in patient's assessment of arthritis pain according to visual analogue scale | Week 6

SECONDARY OUTCOMES:
Change from baseline in American Pain Society Modified Brief Pain Inventory Short Form pain scores | Days 1-7
Change from baseline in patient's assessment of arthritis pain according to visual analogue scale | Week 2
Change from baseline in patient and physician global assessments of arthritis | Weeks 2 and 6
Change from baseline in Western Ontario and McMaster Universities Osteoarthritis Index | Week 6
The Pain Satisfaction Scale | Week 6
The Patient Health Questionnaire (PHQ-9) | Week 6
Measurement of upper gastrointestinal tolerability | Weeks 2 and 6
Adverse events | Weeks 2 and 6
Laboratory test results | Week 6
Vital signs | Weeks 2 and 6
Physical examination | Week 6

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (26):
- Germany (8):
  - Pfizer Investigational Site, Bad Münder am Deister
  - Pfizer Investigational Site, Beckum
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Ostseebad Damp
  - Pfizer Investigational Site, Schwerin
  - Pfizer Investigational Site, Stade
  - Pfizer Investigational Site, Tostedt
  - Pfizer Investigational Site, Weener
- Spain (7):
  - Pfizer Investigational Site, Barcelona
  - Pfizer Investigational Site, Cadiz
  - Pfizer Investigational Site, Guadalajara
  - Pfizer Investigational Site, Madrid
  - Pfizer Investigational Site, Oviedo
  - Pfizer Investigational Site, Seville
  - Pfizer Investigational Site, Valencia
- United Kingdom (11):
  - Pfizer Investigational Site, Chelmsly WOOD, Birmingham
  - Pfizer Investigational Site, Truro, Cornwall
  - Pfizer Investigational Site, Chorley, Lancs
  - Pfizer Investigational Site, Liverpool, Lancs
  - Pfizer Investigational Site, Cannock, Mid Staffordshire
  - Pfizer Investigational Site, Addlestone, Surrey
  - Pfizer Investigational Site, Huddersfield
  - Pfizer Investigational Site, London
  - Pfizer Investigational Site, Manchester
  - Pfizer Investigational Site, Newcastle upon Tyne
  - Pfizer Investigational Site, Wigan

REFERENCES:
- [Derived] Gordo AC, Walker C, Armada B, Zhou D. Efficacy of celecoxib versus ibuprofen for the treatment of patients with osteoarthritis of the knee: A randomized double-blind, non-inferiority trial. J Int Med Res. 2017 Feb;45(1):59-74. doi: 10.1177/0300060516673707. Epub 2017 Jan 12. PMID 28222627
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3191062&StudyName=Efficacy%20and%20Safety%20of%20Celecoxib%20versus%20Ibuprofen%20in%20the%20Treatment%20of%20Osteoarthritis%20of%20the%20Knee%20%28Europe%29